CLINICAL TRIAL: NCT03010930
Title: Does Repeated Dietary Exposure to Umami Taste Affect Umami Perception, Hedonics, or Satiety? A Randomized Controlled Study
Brief Title: Repeated Exposure to Umami Taste on Taste Perception, Hedonics, and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1608006563
Record Dates: First submitted 2016-12-15; First posted 2017-01-05 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Umami Taste Perception
MeSH Terms: interventions — Sodium Glutamate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increased exposure to MSG (Experimental): Subjects consume vegetable broth daily containing MSG
  Interventions: Other: Supplementation of diet with MSG
- No change in exposure to MSG (Sham Comparator): Subjects consume low glutamate vegetable broth daily, sodium-matched to the broth of the experimental group with NaCl
  Interventions: Other: No supplementation of diet with MSG

INTERVENTIONS:
Other: Supplementation of diet with MSG — Subjects eat normal diet and consume 8 ounces of vegetable broth with added MSG one time per day for 1 month
  Arms: Increased exposure to MSG
Other: No supplementation of diet with MSG — Subjects eat normal diet and consume 8 ounces of low glutamate vegetable broth without MSG (sodium-matched with NaCl) one time per day for 1 month
  Arms: No change in exposure to MSG

SUMMARY:
The purpose of this study is to determine how repeated dietary exposure to umami taste affects umami taste perception, hedonics, food preferences, and satiety. Healthy adult subjects will consume a low glutamate vegetable broth daily for one month, where the experimental group's broth is supplemented with the umami-rich stimuli of monosodium glutamate (MSG) and the control group's low glutamate broth is matched for sodium (NaCl).

The investigators hypothesize that repeated dietary exposure to umami taste will:

1. diminish umami suprathreshold intensity perception and hinder the ability to discriminate varying MSG concentrations
2. decrease liking of umami-rich foods and shift preferences upwards towards more intense umami stimuli
3. decrease satiation and decrease the satiating effect of a test meal

ELIGIBILITY:
Inclusion Criteria:

* Have normal sense of taste and smell (self-report)
* Likes soups or broths (self-report)
* Able to report to study site daily (self-report)

Exclusion Criteria:

* Restrained eater (score > 12 on restrained eating subscale from Three Factor Eating Questionnaire)
* BMI < 18 or > 25 kg/m2 (self-report)
* Vegan (self-report)
* Hypertensive or on low-sodium diet (self-report)
* Allergic or sensitive to MSG (self-report)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in umami taste intensity perception | 1 month (at baseline and post intervention)
  Subjects rate the umami intensity of aqueous solutions and foods on the general Labeled Magnitude Scale before and after a month-long dietary supplementation to determine how perception changes with repeated exposure to umami taste
Change in umami taste discrimination | 1 month (at baseline and post intervention)
  Subjects rank solutions of varying umami intensity before and after a month-long dietary supplementation to determine how perception changes with repeated exposure to umami taste

SECONDARY OUTCOMES:
Change in umami liking and preference | 1 month (at baseline and post intervention)
  Subjects rate liking and preference in a variety of umami-rich foods before and after a month-long dietary supplementation to determine how liking and preference of umami-rich foods changes with repeated exposure to umami taste
Change in liking and wanting of high protein foods | 1 month (at baseline and post intervention)
  Subjects complete the Leeds Food Preference Questionnaire before and after a month-long dietary supplementation to determine how explicit liking and implicit wanting of high-protein foods changes with repeated exposure to umami taste
Change in satiation | 1 month (at baseline and post intervention)
  Subjects consume a test meal and the amount of food eaten is measured before and after a month-long dietary supplementation to determine how satiation from a test meal differs after repeated exposure to umami taste
Change in satiety | 1 month (at baseline and post intervention)
  Subjects consume a test meal and rate appetite sensations on a visual analog scale throughout the test meal before and after a month-long dietary supplementation. A satiety quotient will be derived from these values with the formula: Satiety Quotient = (rating pre-eating episode-rating post-eating episode) / (intake of eating episode) to determine how satiety changes with repeated exposure to umami taste

OTHER OUTCOMES:
Height | 1 month (at baseline and post intervention)
  Body height (centimeters) will be measured with standard procedures and equipment. Using this information, BMI will be calculated with the formula: BMI=[kg/m]2 to ensure that BMI does not change with repeated exposure to umami taste
Weight | 1 month (at baseline and post intervention)
  Body weight (kilograms) will be measured with standard procedures and equipment. Using this information, BMI will be calculated with the formula: BMI=[kg/m]2 to ensure that BMI does not change with repeated exposure to umami taste
Habitual glutamate consumption | 1 month (at baseline and post intervention)
  Subjects complete the National Cancer Institute's monthly diet history questionnaire to estimate habitual glutamate consumption. Baseline habitual glutamate consumption, in addition to gender, will be assessed as effect modifiers in the analysis.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noel CA, Finlayson G, Dando R. Prolonged Exposure to Monosodium Glutamate in Healthy Young Adults Decreases Perceived Umami Taste and Diminishes Appetite for Savory Foods. J Nutr. 2018 Jun 1;148(6):980-988. doi: 10.1093/jn/nxy055. PMID 29796671